CLINICAL TRIAL: NCT02391792
Title: Membrane Shedding During Severe Sepsis and Septic Shock: Pathophysiological and Clinical Relevance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: DC2012-1633
Record Dates: First submitted 2014-09-04; First posted 2015-03-18 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Severe Sepsis and Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients: patients with septic shock
- control: patients without septic shock
- healthy volunteers

SUMMARY:
Microparticules (MPs) result from plasma cell membrane remodeling and shedding after cell stimulation or apoptosis. MPs are know recognized as a pool of bioactive messengers with merging role in pathophysiology of immune and cardiovascular diseases. MPs have been characterized during septic shock and may contribute to dissemination of pro-inflammatory and procoagulant mediators. This a prospective observational study of circulating MPs and blood coagulation in septic shock patients admitted in medical intensive care units (ICUs) of four tertiary hospitals at baseline (D1, D2, D3, D4, D7).

ELIGIBILITY:
Inclusion Criteria:

* Septic shock (patients)
* Without septic shock (control)
* Informed consent

Exclusion Criteria:

* Class IV heart failure
* Child-plugh grade C cirrhosis
* Cancer under active treatment
* BMI>35kg/m2
* Moribund patient
* DNR decision

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: group patient: patients with septic shock group control: patients without septic shock
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-03; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in number and type of circulating microparticles at 7 days | Baseline and 7 days
Change from baseline in blood coagulation markers at 7 days | Baseline and 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nouvel Hopital Civil, Strasbourg, Alsace, France

REFERENCES:
- [Derived] Helms J, Severac F, Merdji H, Clere-Jehl R, Francois B, Mercier E, Quenot JP, Meziani F; CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). Performances of disseminated intravascular coagulation scoring systems in septic shock patients. Ann Intensive Care. 2020 Jul 10;10(1):92. doi: 10.1186/s13613-020-00704-5. PMID 32651674